CLINICAL TRIAL: NCT06940492
Title: A Mediation Analysis Investigating Dry Needling Treatment Mechanisms in a Chronic Low Back Pain Population
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB202500403
Record Dates: First submitted 2025-04-07; First posted 2025-04-23 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-04

CONDITIONS: Chronic Low Back Pain (CLBP)
Keywords: low back pain; chronic low back pain; dry needling
MeSH Terms: conditions — Low Back Pain | interventions — Dry Needling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Dry needling (Experimental): The participant will be placed prone. The skin on each side of the spine at the level of the identified trigger point will be prepped and cleaned with an alcohol swab. Four 50mm - 60 mm filiform needles will be used to penetrate the skin in the lower back; two needles will be inserted bilaterally on each side of the spine at the level of the trigger point. Needles will be placed approximately 1.5cm lateral to the spinous process, directed at a 20 to 30-degree inferior medial angle into the lumbar multifidus. Needles will be manipulated with an "in and out" pistoning technique for 5 - 10 seconds when first inserted into the muscle. After 5 -10 second , the needles will be left resting in the muscle for 10 minutes. Participants will receive 3 sessions of dry needling. Each session will be approximately 72-96 hours apart.
  Interventions: Other: Dry needling

INTERVENTIONS:
Other: Dry needling — Dry needling is a force-based manipulation technique used by health care providers. Force-based manipulation describes when forces external to the body are passively applied to tissue with a therapeutic intent. During dry needling, a filiform needle (i.e., one without medication) is inserted into a muscle to target a trigger point, often times with the intent of eliciting a localized twitch response

SUMMARY:
Low back pain is a common problem that many adults experience at some point in their lives. One treatment being studied is dry needling, a technique where a small needle is inserted into a specific area of muscle to help relieve pain. So far, the research on dry needling for low back pain hasn't been clear, and it's hard to know when and for whom it will work best. This study aims to figure out how dry needling works to help people with chronic low back pain by looking at the underlying factors. By understanding how dry needling helps people, we can develop a more targeted approach to treatment, which could lead to better outcomes for people with chronic low back pain. The goal of this study is to identify the factors that make dry needling effective for people with chronic low back pain, so that this this information can be used to provide more personalized and effective care.

Eligible participants will attend 5 research sessions lasting approximately 1 hour and complete 2 online surveys. At 3 of those sessions, participants will receive dry needling to their low back.

As part of the research, participants will complete questionnaires related to how pain effects their life. Participants will also undergo testing for muscle stiffness, low back mobility and strength, and pain sensitivity.

To be included in this study participants must:

* Be 18-65 years of age
* Have low back pain for at least 3 months

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18 - 65,
2. Currently experiencing pain in the space between the twelfth rib and the horizontal gluteal fold with or without radiating leg pain

b) Low back pain symptoms that are chronic, in that symptoms, have persisted for at least 3 months with pain experienced on most or every day in the past 3 months c) Not currently receiving treatment for their low back

Exclusion Criteria:

1. Non-English speaker
2. presence of a medical condition known to affect sensation
3. history of surgery to the low back
4. history of blood clotting disorders or medical conditions associated with bleeding disorders
5. Current use of the medication causing difficulty with clotting (such as blood thinners)
6. Contraindication to the application of needles including, but not limited to, diabetes, local infection, epilepsy, fear of needles or metal allergy
7. women who are pregnant or currently attempting to become pregnant
8. diagnosis of active cancer
9. inability to obtain the testing position (laying prone).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Will be collected at the baseline visit, seventy-two hour follow up, and at 2- and 4-week follow up. Current pain intensity will also be assessed at each dry needling session immediately before and immediately after receiving the intervention
  Pain intensity will be assessed using the Brief Pain Inventory's (BPI) pain intensity sub-scale. The BPI pain intensity sub-scale creates an average score of pain intensity by assessing four pain intensity domains of the current, best, and worst pain in the past twenty-four hours and pain on average, then adding these scores together and taking an average. The pain intensity domains are measured using the numeric pain rating scale (NPRS) anchored at "0" (no pain) and "10" (The worst pain imaginable).

SECONDARY OUTCOMES:
Patient Reported Outcomes Measurement Inventory System version 2.0(PROMIS-29) | PROMIS 29 subscales will be measured at baseline, at the needling session following the baseline visit, seventy-two hour follow up, and 2 and 4 week follow up
  The PROMIS-29 is a National Institute of Health-supported outcome measure that assesses multiple domains, including pain intensity with the NPRS an average of pain in the past seven days, physical function, fatigue, pain interference, ability to participate in social roles and activity, symptoms of anxiety, symptoms of depression, and sleep disturbance

OTHER OUTCOMES:
The Participant Global Impression of Change (PGIC) | The PGIC will be administered at seventy-two-hour, two-week, and four-week follow-ups
  The PGIC is a single-item, seven-point measure ranging from "Very much improved" to "Very much worse" and is responsive to change in chronic pain samples
The Physical Impairment Index (PII) | The PII will be administered at the baseline session, at each of the 3 dry needling sessions immediately before and immediately after receiving the intervention, and seventy-two-hour follow-up
  The PII is a seven-item test of various ranges of motion (ROM) and strength measures specific to the low back. These seven tests include total flexion ROM, total extension ROM, average lateral flexion ROM, average straight leg raise ROM, spinal tenderness, bilateral active straight leg raise, and active sit-up. Each test is scored as a positive or negative, resulting in a "1" or "0" score for a total possible score of seven. A higher score indicates higher levels of impairment
Myotonometry | Myotonometry collection will occur at the baseline session, at each of the 3 needling session immediately before and immediately after receiving the intervention, and seventy-two-hour follow-up
  Myotonometry measures global soft tissue biomechanical and viscoelastic properties. Myotonometry can be performed with handheld devices to quantify soft tissue properties. the MyotonPro handheld device will be used to collect myotonometry measurements. For this investigation, the MyotonPro (MyotonPro, Myoton Ltd.s., Tallinn, Estonia) will be used to collect myotonometry measurements of dynamic stiffness. The measure of dynamic stiffness is a measure of soft tissue resistance to deformation of its initial shape in response to internal or external forces. The measure of stiffness in newtons per meter will be collected at the spinal level of L4 on the side of the most tender trigger point
Pressure pain threshold | Pressure pain threshold measures will be collected at the baseline session, at each of the 3 needling session immediately before and immediately after receiving the intervention, and at seventy-two-hour follow-up
  Pressure pain threshold testing will be measured at the lower back just medial to the posterior superior iliac spine (PSIS) and on the proximal anterior tibialis (approximately 5cm from Girdy's Tubercle) on the side of the most tender trigger point. Threshold testing will be performed using a digital pressure algometer (Wagner Instruments FPX 25, Greenwich, CT) with a 1 cm diameter rubber tip with pressure applied perpendicular to the testing area at a rate of 1 kgf/s. Participants will be instructed to verbally indicate when the sensation first changed from pressure to pain and the amount of pain intensity with the NPRS. The NPRS will be anchored at "0" (no pain) and "100" (The worst pain imaginable). Pressure pain threshold testing will be performed two times, with an average of the two measures used for analysis.
Pain catastrophizing scale (PCS) | The PCS will be collected at the dry needling session number 1 (the session following the baseline session) and seventy-two-hour follow-up
  The PCS is a thirteen-item questionnaire in which participants rate each item from 0 to 4, with larger numbers indicating higher levels of pain catastrophizing. The PCS is extensively studied as an assessment of pain catastrophizing and has sound psychometric properties.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No